CLINICAL TRIAL: NCT02676882
Title: EnBrace HR for Depression Treatment and Prevention in Women Trying to Conceive and Early Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: JayMac Pharmaceuticals, LLC (Unknown)
Responsible Party: Principal Investigator, Marlene P. Freeman, MD, Associate Director, Center for Women's Mental Health, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016P000275
Record Dates: First submitted 2016-02-04; First posted 2016-02-08 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Depressive Disorder; Pregnancy
Keywords: Depressive Disorder; Depression; Antidepressants; Pregnancy; Folate; Dietary Supplements; Omega-3 Fatty Acids; Women's Health; Vitamins
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Intervention Model Description: A pilot study of EnBrace HR in two groups of women with major depressive disorder (MDD). Group 1 includes women who are well at time of enrollment and are not experiencing clinically significant depressive symptoms. In this group, EnBrace HR is studied for depressive relapse prevention during the perinatal period. Group 2 includes women who are depressed at time of enrollment and who are currently experiencing clinically significant depressive symptoms. In this group, EnBrace HR is assessed for acute treatment of MDD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EnBrace HR for Prevention of Depressive Relapse (Group 1) (Other): Prescription folate prenatal supplement with other dietary ingredients; one multiphasic soft gelatin capsule 1x/day for 12 weeks. Participants are not currently in a depressive episode per the Mini International Neuropsychiatric Interview (MINI) and are not experiencing clinically significant depression symptoms assessed using the Montgomery Asberg Depression Rating Scale (MADRS) with a score </= 10.
  Interventions: Dietary Supplement: EnBrace HR
- EnBrace HR for Acute Treatment of Major Depression (Group 2) (Other): Prescription folate prenatal supplement with other dietary ingredients; one multiphasic soft gelatin capsule 1x/day for 12 weeks. Participants are currently in a depressive episode per the Mini International Neuropsychiatric Interview (MINI) and are experiencing clinically significant depression symptoms assessed using the Montgomery Asberg Depression Rating Scale (MADRS) with a score >/= 15.
  Interventions: Dietary Supplement: EnBrace HR

INTERVENTIONS:
Dietary Supplement: EnBrace HR — Prescription folate prenatal supplement with other dietary ingredients; one multiphasic soft gelatin capsule 1x/day for 12 week study

SUMMARY:
The purpose of this study is to assess the effectiveness of the EnBrace HR prenatal supplement in preventing depression in women with a history of depression who have decided to stop taking antidepressants during their pregnancy, or treating women who are currently in a depressive episode while pregnant or planning pregnancy.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) occurs twice as often in women as in men, with an age of onset that coincides with the childbearing years. As over 20% of reproductive-age women experience an episode of depression, identifying safe and effective treatments for depression before, during and after pregnancy has become a critical public health issue. Historically, pregnancy has been viewed as a protective time with respect to risk for psychiatric illnesses, which has resulted in a lack of prospective systematic investigations on the subject of acute treatment and prevention of MDD while women are planning to conceive and during pregnancy. Contrary to previous assumptions, recent large-scale studies demonstrate that new onset and recurrence of depressive episodes occur commonly during pregnancy and the postpartum periods. The current standard of treatment for recurrent major depression is maintenance antidepressant (AD) therapy, due to the high risk of recurrence among patients who discontinue maintenance AD therapy.

Although ADs are frequently used during pregnancy, concerns remain regarding a spectrum of adverse outcomes associated with fetal exposure to these medications including: increased risk for teratogenicity compromised obstetrical outcomes and a variety of negative neonatal clinical syndromes. Given these concerns, reproductive age women treated with AD frequently elect to discontinue their medications proximate to pregnancy or immediately after becoming pregnant despite the known increased risk for relapse or recurrence. With the exception of observational data that demonstrate that women who discontinue medication around the time of conception are at high risk of recurrence, no previous studies are available to inform clinical treatment regarding medication discontinuation for a planned pregnancy.

This leaves women who are successfully treated with ADs and want to become pregnant caught in the difficult clinical dilemma of weighing the risks of fetal exposure to medication against the potential impact of untreated maternal depression during pregnancy. Clinical decisions are made even more complex by the fact that most studies are far from definitive in terms of comparing the risks of in utero exposure to ADs to the risks of untreated antenatal mood disorder. Given this level of uncertainty, many women and their health care providers would welcome evidence-based non-psychotropic interventions as an alternative to ADs in order to prevent recurrence in euthymic women with histories of MDD as they plan pregnancy. However, the potential efficacy of non-psychotropic interventions for this population has not been systematically investigated.

There is consistent and growing evidence of a role for various folate forms in the prevention and treatment of depression. In fact, there is compelling evidence that treatment with a methylfolate agent would not only avoid the potential risks of antidepressants in pregnancy, but would also confer important benefits to pregnancy and child outcomes as well, such as prevention of major birth defects and longer term neurodevelopmental outcomes. To date, there is an evidence base for antidepressant effects for folic acid, folinic acid, and methylfolate, and similar findings may be attributable to the fact that these folate forms share an interconversion potential in the complex set of pathways that comprise the one-carbon cycle. These reactions, which in turn depend on B12 and homocysteine availability, are postulated to exert an antidepressant effect by impacting the synthesis of neurotransmitters such as norepinephrine, dopamine, and serotonin.

Some but not all studies suggest efficacy of folate monotherapy for MDD, but this intervention may be limited by the common occurence of polymorphisms in the general population that make folate a less efficient one-carbon cycle constituent than L-methylfolate. Since certain polymorphisms that impair methylation processes and the conversion of folate into its active form, methylfolate, have been found to be overrepresented in individuals with depression, methylfolate may be a more effective form of folate supplementation to target MDD. Also, methylfolate may be more readily absorbed in the brain compared to other folate forms.

Recently, Fava and colleagues demonstrated that L-methylfolate is significantly superior to placebo for the treatment of major depressive disorder in patients who had failed to respond to AD therapy alone. In addition, several other open and blinded studies of methylfolate monotherapy in a variety of depressed populations have found that patients experienced significant improvement in depressive symptoms with no drug-related adverse events. Although more controlled data are needed, initial studies indicate that methylfolate may be a safe and effective option for the treatment of depression, especially in populations that are vulnerable to medication-related adverse events, and those who are folate deficient or whose folate needs are elevated, such as the case in pregnant women.

EnBrace HR is a prescription prenatal/postnatal dietary management product that contains vitamins and minerals, including folic acid and methylfolate. It meets the above criteria as a potential ideal candidate for the prevention of depression in pregnancy. It contains L-methylfolate and other folate derivatives, and is optimal for a population with high rates of polymorphisms that affect folic acid metabolism. It also contains omega-3 fatty acids, primarily eicosapentaenoic acid, which shows promise for the treatment of depression. Importantly, these components are crucial for healthy pregnancies. Folic acid supplementation has been associated with the reduced risk of neural tube defects and is recommended for use in women of reproductive potential to reduce the risk of birth defects, although a substantial proportion of the population are poor folic acid metabolizers. Methylfolate compounds specifically may provide a more efficient delivery of folate-related compounds to this end.

Very few studies have examined treatments specifically to assist patients that discontinue ADs, and none have examined this during the time proximate to attempts to conceive, or during pregnancy, which is particularly relevant due to safety concerns. The adaptation of a non-psychotropic treatment, such as EnBrace, for use in women who are planning pregnancy or who are pregnant who choose to discontinue maintenance AD treatment would broaden treatment choices available during this important time in the female life-cycle.

Objective: The overarching goal of this investigation is to assess EnBrace as a treatment for the acute treatment and prevention of depression in women with a history of major depressive disorder who decide to avoid or discontinue their maintenance AD treatment for pregnancy. After completing this protocol, we plan to use the preliminary data for the development of a randomized controlled trial protocol. We will include two groups of women who are interested in minimizing medication exposures while trying to conceive or during pregnancy: 1) women who have histories of depression and are not depressed, and would like to stop antidepressants for pregnancy, 2) women in depressive episodes who are pregnant or trying to conceive (on or off of antidepressant medications).

Specific Aim 1a: To evaluate the efficacy of EnBrace when used as maintenance treatment for MDD in a group of women (N=10) who are trying to conceive or are early in pregnancy and who have decided to stop ADs (Group 1). Relapse rates for women in this context have been demonstrated to be high, with 68% relapse rates in a large multisite NIMH-funded trial.

Specific Aim 1b: To evaluate the efficacy of EnBrace when used as an acute treatment for MDD in a group of women (N=10) who are trying to conceive or are early in pregnancy (Group 2). Women will have major depressive episodes in this group, and may receive EnBrace as monotherapy, or as an adjunct to current pharmacotherapy.

Hypothesis 1a: We hypothesize that relapse rates will be lower for women who receive EnBrace compared to historical controls. MDD relapse will be determined by the Mini-International Neuropsychiatric Interview (MINI) mood module that will be administered by a study clinician at each visit.

Hypothesis 1b: We hypothesize that the majority of women who receive EnBrace will experience a response (50% improvement in depressive symptoms) to EnBrace therapy.

Specific Aim 2: To identify biological markers as potential predictors of response to EnBrace.

Hypothesis 2: We hypothesize that pre- to post-treatment changes in homocysteine, folate, B12, IL-6 and CRP will be associated with response to EnBrace. We hypothesize specifically that levels of folate and B12 will increase and homocysteine will decrease temporally with treatment and be predictive of prevention of depressive episodes. We hypothesize that treatment will lower IL-6 and CRP levels due to the anti-inflammatory components of EnBrace (i.e., omega-3 fatty acids) and that decreased levels of inflammatory markers may predict lower risk of depressive relapse in participants who enter the study while not on a depressive episode (Group 1), and will predict response to treatment in women who enter the study while in a depressive episode (Group 2).

Specific Aim 3 (Exploratory): To identify factors influencing adherence to and tolerability of treatment. This will be achieved by using qualitative methods to explore (a) perceived risks and benefits of treatment; (b) perceived side effect profile; (c) treatment convenience; (d) knowledge of, attitudes towards, and preferences for depression treatment while attempting to conceive or early pregnancy.

Hypothesis 3: We hypothesize that EnBrace will be perceived by patients as 1) an acceptable and attractive treatment with a favorable risk/benefit profile in the context of pregnancy or while trying to conceive, 2) well tolerated, 3) convenient and easy to adhere to, 4) will be a treatment that women who are trying to conceive or who are pregnant find intuitive and preferable to prescription antidepressant medication (or for women on antidepressant treatment in Group 2, who prefer the augmentation with EnBrace rather than an increase in antidepressant dose or augmentation with a prescription psychotropic medication).

ELIGIBILITY:
Inclusion Criteria:

Group 1 (Observational, not-randomized)

Inclusion Criteria:

1. Planning pregnancy or pregnant < 28 weeks gestation
2. Currently meet criteria for stable remission from MDD, defined as a baseline score of < 10 on the Montgomery-Åsberg Depression Rating Scale (MADRS)
3. Current or recent treatment with an AD
4. Have elected to discontinue AD medication for pregnancy (may have already begun or completed taper)
5. Have a history of a major depressive episode/ Previous Episode of MDD, as verified using the MINI Structured Clinical Interview for DSM-5; have MDD as one of their primary diagnoses
6. Has a treating prescribing clinician for the treatment of MDD

Exclusion Criteria:

1. Current major depressive episode, as diagnosed on the MINI mood portion
2. Significant risk for self-harm or harm to others
3. Psychotic symptoms
4. Meeting criteria for a primary diagnosis of schizophrenia, an active eating disorder, dementia, delirium, or other cognitive disorder
5. Presence of an active substance and/or alcohol abuse disorder within six months prior to screening
6. Pernicious anemia or history of gastric bypass surgery
7. Seizure disorder and/or on anticonvulsant medications
8. Allergy to beeswax, soy, fish, nuts, peanuts, egg, wheat, milk, and/or shellfish
9. Non-English speaking

Group 2

Inclusion Criteria:

1. Planning pregnancy or pregnant < 28 weeks gestation
2. Currently experiencing clinically significant depressive symptoms, defined as a baseline score of > 15 on the Montgomery-Åsberg Depression Rating Scale (MADRS)
3. Experiencing a major depressive episode, as verified using the MINI Structured Clinical Interview for DSM-5; have MDD as one of their primary diagnoses
4. Has a treating prescribing clinician for the treatment of MDD

Exclusion Criteria:

1. Significant risk for self-harm or harm to others
2. Psychotic symptoms
3. Meeting criteria for a primary diagnosis of schizophrenia, an active eating disorder, dementia, delirium, or other cognitive disorder
4. Presence of an active substance and/or alcohol abuse disorder within six months prior to screening
5. Pernicious anemia or history of gastric bypass surgery
6. Seizure disorder and/or on anticonvulsant medications
7. Allergy to beeswax, soy, fish, nuts, peanuts, egg, wheat, milk, and/or shellfish
8. Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene P Freeman, MD, Principal Investigator — Massachusetts General Hospital, Center for Women's Mental Health
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
All data will be presented in aggregate to protect participant privacy.

REFERENCES:
- [Result] Cohen LS, Altshuler LL, Harlow BL, Nonacs R, Newport DJ, Viguera AC, Suri R, Burt VK, Hendrick V, Reminick AM, Loughead A, Vitonis AF, Stowe ZN. Relapse of major depression during pregnancy in women who maintain or discontinue antidepressant treatment. JAMA. 2006 Feb 1;295(5):499-507. doi: 10.1001/jama.295.5.499. PMID 16449615

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 1/24/2017 through 3/5/2018 Recruitment methods: Medical clinics, womensmentalhealth.org, other online recruitment sources, flyers in public locations, database of previous patients and research participants at the Center for Women's Mental Health at MGH
Pre-assignment Details: Potential subjects were screened by phone and if eligible attended a baseline screening visit at which they consented to further eligibility assessment for each of two groups. If after consent they failed to meet eligibility criteria, they were considered enrolled per IRB guidelines, but were not assigned to a group to start study medication.
Groups:
- Group 1 - Relapse-Prevention Group ("Well" Group): Inclusion criteria: women ages 18+ who currently meet criteria for stable remission from MDD as defined by a baseline score of < 10 on the Montgomery-Åsberg Depression Rating Scale (MADRS),have recent or current antidepressant use which they have elected to discontinue for pregnancy, have histories of an MDE as verified using the Mini-International Neuropsychiatric Interview (MINI) for DSM-IV, and have MDD as one of their primary diagnoses.
  Treatment: EnBrace HR, a prescription folate prenatal supplement with other dietary ingredients; one multiphasic soft gelatin capsule 1x/day for 12 week study
- Group 2 - Treatment Group ("Depressed" Group): Inclusion criteria: Women ages 18+ who are currently experiencing clinically significant depressive symptoms as defined by a baseline score of > 15 on the MADRS, planning not to start an antidepressant or to increase the dose of a current antidepressant after consultation with their prescribing provider, currently experiencing an MDE as verified using the MINI, and have MDD as one of their primary diagnoses. Women who endorsed any suicidal ideation were not included in the study, and follow-up care was swiftly coordinated.
  Treatment: EnBrace HR, a prescription folate prenatal supplement with other dietary ingredients; one multiphasic soft gelatin capsule 1x/day for 12 week study
Period: Overall Study
Arm/Group | Group 1 - Relapse-Prevention Group ("Well" Group) | Group 2 - Treatment Group ("Depressed" Group)
Started | 13 | 7
Evaluable (Received study drug; completed minimum 1 follow-up visit; if Group 1, discontinued antidepressants.) | 11 | 6
Completed | 10 | 5
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Relapse-Prevention Group ("Well" Group) | Group 2 - Treatment Group ("Depressed" Group) | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 7 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 32.2 [28 to 35] | 35.3 [31 to 39] | 32.8 [28 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 13 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 5 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 7 | 20
Mini International Neuropsychiatric Interview Major Depressive Episode Module [Count of Participants; unit: Participants] — A brief, validated structured clinical interview used for diagnostic purposes for DSM-IV and ICD-10 psychiatric disorders in clinical trials. The interview is performed by a licensed study physician and takes about 15 minutes. The MINI is divided into modules corresponding to diagnostic categories, and questions are answered as a binary yes or no by the research subject. The MINI mood module in this case refers to the set of questions examining major depressive disorder symptoms to identify if a patient is experiencing depressive symptoms that meet criteria as a major depressive episode.
  Participants | 0 | 7 | 7
Montgomery-Asberg Depression Rating Scale (MADRS) Score </= 10 [Count of Participants; unit: Participants] — A 10-item scale assessing the presence and severity of depressive symptoms, each with a score of 0-6 in which 0 denotes absence of a given symptom and 6 denotes the highest burden, frequency, or severity of a given symptom. The total score (sum of 10 items) ranges from 0-60 points, with scores of </=10 considered clinically well and scores of >/=15 considered clinically depressed for this study. Symptoms assessed include reported and apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulty, lassitude, anhedonia, pessimistic thoughts, and suicidality.
  Participants | 13 | 0 | 13
Montgomery-Asberg Depression Rating Scale (MADRS) >/= 15 [Count of Participants; unit: Participants] — A 10-item scale assessing the presence and severity of depressive symptoms, each with a score of 0-6 in which 0 denotes absence of a given symptom and 6 denotes the highest burden, frequency, or severity of a given symptom. The total score (sum of 10 items) ranges from 0-60 points, with scores of </=10 considered clinically well and scores of >/=15 considered clinically depressed for this study. Symptoms assessed include reported and apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulty, lassitude, anhedonia, pessimistic thoughts, and suicidality.
  Participants | 0 | 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in the Relapse-Prevention Group (Group 1) Experiencing a Major Depressive Episode Relapse
Description: Evidence of recurrence of major depression episode, as defined by the Mini-International Neuropsychiatric Interview (MINI) mood module and/or research clinician interview. The MINI is a brief, validated structured clinical interview used for diagnostic purposes for DSM-IV and ICD-10 psychiatric disorders in clinical trials. The interview is performed by a licensed study physician and takes about 15 minutes. The MINI is divided into modules corresponding to diagnostic categories, and questions are answered as a binary yes or no by the research subject. The MINI mood module in this case refers to the set of questions examining major depressive disorder symptoms to identify if a patient is experiencing depressive symptoms that meet criteria as a major depressive episode.
Time Frame: Assessed every two weeks for 12 weeks
Population: Those women in group 1 who discontinued antidepressants (ADs) during the study (2 women of 13 in group 1 planned to discontinue ADs when they became pregnant and were actively trying to conceive, but they did not become pregnant during the trial and did not decrease the dose of their ADs).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Relapse-Prevention Group ("Well" Group)
Number analyzed (Participants) | 11
Participants | 3
Statistical Analysis 1: Comparison: Group 1 - Relapse-Prevention Group ("Well" Group); Test type: Other — A Chi Squared analysis was performed to determine how the rate of relapse in Group 1 (27.3%) compared to that of historical controls in the literature (67.7%). (Cohen, JAMA 2006); p = 0.005, Chi-squared — A priori threshold for statistical significance: p<0.05

2. Primary Outcome: Rate of Treatment Response Among Depressed Participants (Group 2) to EnBrace Therapy Measured Using the Montgomery Asberg Depression Rating Scale
Description: Experience a response (50% improvement in depressive symptoms) to EnBrace therapy, as assessed by the Montgomery Asberg Depression Rating Scale (MADRS). The MADRS is a 10-item scale assessing the presence and severity of depressive symptoms, each with a score of 0-6 in which 0 denotes absence of a given symptom and 6 denotes the highest burden, frequency, or severity of a given symptom. The total score (sum of 10 items) ranges from 0-60 points, with scores of </=10 considered clinically well and scores of >/=15 considered clinically depressed for this study. Symptoms assessed include reported and apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulty, lassitude, anhedonia, pessimistic thoughts, and suicidality.
Time Frame: Assessed every two weeks for 12 weeks
Population: Of the 7 women eligible for inclusion in Group 2, 1 did not initiate study medication and dropped from the study after baseline. The 6 other women were evaluable as they returned for follow-up visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 - Treatment Group ("Depressed" Group)
Number analyzed (Participants) | 6
Participants | 5
Statistical Analysis 1: Comparison: Group 2 - Treatment Group ("Depressed" Group); Test type: Other — A one-way repeated measures ANOVA was used to examine the overall course of Group 2 participants' MADRS scores. (F(6, 29)=5.16, p=0.001); p = 0.001, ANOVA — a priori threshold for statistical significance: p <0.05

ADVERSE EVENTS:
Time Frame: Participants were followed for up to 9 months - 3 months in the treatment phase and 6 months in the optional follow-up phase.
Description: Adverse event information was collected at each visit using a standardized adverse event reporting form and assessed by a licensed physician for severity. If a participant could not report to a visit due to a serious adverse event, this information was also recorded. If a participant was not exposed to the study medication, they were not included in the total number of participants at risk. This occurred in Group 2, in which 1 participant dropped from the study prior to medication initiation.
Groups:
- Group 1 - Relapse Prevention Group ("Well" Group): Treatment: EnBrace HR - prescription folate prenatal supplement with dietary ingredients; one multiphasic gelatin capsule/day for 12 weeks.
  Inclusion criteria: women ages 18+ who currently meet criteria for stable remission from Major Depressive Disorder (MDD) as defined by a baseline score of </=10 on the Montgomery-Åsberg Depression Rating Scale (MADRS), have recent or current antidepressant use which they have elected to discontinue for pregnancy, have histories of a major depressive episode (MDE) as verified using the Mini-International Neuropsychiatric Interview (MINI) for DSM-IV, and have MDD as one of their primary diagnoses.
- Group 2 - Treatment Group ("Depressed" Group): Treatment: EnBrace HR - prescription folate prenatal supplement with dietary ingredients; one multiphasic gelatin capsule/day for 12 weeks.
  Inclusion criteria: Women ages 18+ who are currently experiencing clinically significant depressive symptoms as defined by a baseline score of >/=15 on the MADRS, planning not to start an antidepressant or to increase the dose of a current antidepressant after consultation with their prescribing provider, currently experiencing an MDE as verified using the MINI, and have MDD as one of their primary diagnoses. Women who endorsed any suicidal ideation were not included in the study, and follow-up care was swiftly coordinated.
Arm/Group | Group 1 - Relapse Prevention Group ("Well" Group) | Group 2 - Treatment Group ("Depressed" Group)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/6
Other Adverse Events (participants affected / at risk) | 10/13 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Relapse Prevention Group ("Well" Group) (N=13) | Group 2 - Treatment Group ("Depressed" Group) (N=6)
major depressive episode requiring inpatient hospitalization (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Relapse Prevention Group ("Well" Group) (N=13) | Group 2 - Treatment Group ("Depressed" Group) (N=6)
Nausea with onset during pregnancy (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Cough and nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Difficulty concentrating (Psychiatric disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal muscle ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Suspected niacin flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mechanical fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mild anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Worsening of depression symptoms with request for treatment referral (Psychiatric disorders) | 0 (0) | 1 (1)
Mild weight gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Chest tightness (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations:

* Lack of a placebo arm
* Small number of subjects in each group and overall
* Over-representation of white, non-Hispanic, married, and highly-educated women

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT02676882/Prot_SAP_000.pdf